CLINICAL TRIAL: NCT01868061
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Lebrikizumab in Patients With Uncontrolled Asthma Who Are on Inhaled Corticosteroids and a Second Controller Medication
Brief Title: A Study of Lebrikizumab in Participants With Uncontrolled Asthma on Inhaled Corticosteroids and a Second Controller Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB28689; 2013-000176-15 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Lebrikizumab (125 mg) (Experimental): Participants will receive SC injection of lebrikizumab (125 mg) every 4 weeks for 104 weeks.
  Interventions: Drug: Lebrikizumab
- Lebrikizumab (37.5 mg) (Experimental): Participants will receive SC injection of lebrikizumab (37.5 mg) every 4 weeks for 104 weeks.
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Participants will receive SC injection of lebrikizumab matching placebo every 4 weeks for 52 weeks during placebo-controlled period and then SC injection of lebrikizumab at 125 or 37.5 mg for 52 weeks during active treatment extension period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered as SC injection at 125 or 37.5 mg every 4 weeks, for 104 weeks.
  Other Names: RO5490255
Drug: Placebo — Lebrikizumab matching placebo will be administered as SC injection every 4 weeks for 52 weeks.
  Arms: Placebo

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of lebrikizumab in participants with asthma whose disease remains uncontrolled despite daily treatment with inhaled corticosteroid (ICS) therapy and at least one second controller medication. Participants will be randomized in 1:1:1 ratio to receive double-blind treatment with either lebrikizumab ("high" or "low") or placebo, administered as subcutaneous (SC) injection every 4 weeks for 52 weeks, in addition to their standard-of-care therapy. This will be followed by a 52-week double-blind active treatment extension. Participants who were assigned to placebo during the placebo-controlled period of the trial will be re-randomized at Week 52 to receive blinded SC lebrikizumab 37.5 milligrams (mg) or 125 mg every 4 weeks from Weeks 53 to 104. The anticipated time on study treatment is 104 weeks. After study treatment, all participants will complete a 20-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis for greater than equal to (>/=) 12 months at Visit 1
* Bronchodilator response at Visit 1, 2, or 3
* Pre-bronchodilator FEV1 of 40 percent (%) - 80% predicted at both Visits 2 and 3
* On ICS therapy at a total daily dose of 500-2000 microgram (mcg) of fluticasone propionate dry powder inhaler (DPI) or equivalent for >/= 6 months prior to Visit 1
* On an eligible second controller medication (long-acting Beta-agonist [LABA], leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonist [LAMA], or theophylline) for 6 months prior to Visit 1
* Uncontrolled asthma at Visit 1 and/or Visit 2, and at Visit 3
* Chest X-ray or computed tomography (CT) scan within 3 months prior to Visit 1 or chest X-ray during the screening period (prior to Visit 3) confirming the absence of other clinically significant lung disease
* Demonstrated adherence with controller medication during the screening period

Exclusion Criteria:

* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Maintenance oral corticosteroid therapy within 3 months of Visit 1
* Treatment with systemic (oral, intravenous [IV], or intramuscular [IM]) corticosteroids within 4 weeks prior to Visit 1 or during the screening period
* Treatment with intra-articular corticosteroids within 4 weeks prior to Visit 1 or during the screening period or anticipated need for intra-articular corticosteroids during the course of the study
* Infection requiring hospital admission for >/=24 hours or requiring treatment with IV or IM antibiotics within 4 weeks prior to Visit 1 or during screening; Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening; Active parasitic infection or Listeria monocytogenes infection within 6 months prior to Visit 1 or during screening
* Active tuberculosis requiring treatment within 12 months prior to Visit 1
* Known immunodeficiency, including, but not limited to, human immunodeficiency virus (HIV) infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* History of interstitial lung disease, chronic obstructive pulmonary disease (COPD), or other clinically significant lung disease other than asthma
* Known current malignancy or current evaluation for potential malignancy
* Current smoker or former smoker with a history of greater than (>) 10 pack-years
* History of alcohol or drug abuse
* Past and/or current use of any anti-interleukin (IL)-13 or anti-IL-4/IL-13 therapy, including lebrikizumab; use of other monoclonal antibody therapy, including omalizumab, within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer) or during screening
* Initiation of or change in allergen immunotherapy within 3 months prior to Visit 1 or during screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1068 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Rate of Asthma Exacerbations During the 52-Week Placebo-Controlled Period | Baseline up to Week 52

SECONDARY OUTCOMES:
Absolute Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) | Baseline, Week 52
Time to First Asthma Exacerbation | Baseline up to Week 52
Change From Baseline in Standardized Asthma Quality of Life Questionnaire (AQLQ) Score | Baseline, Week 52
Change from Baseline In Asthma Rescue Medication (Number of Puffs or Nebulized Treatments) | Baseline, Week 52
Rate of Urgent Asthma-Related Urgent Health Care Utilization | Baseline up to Week 52
Percentage of Participants With Adverse Events | Baseline up to Week 124
Percentage of Participants With Anti-Therapeutic Antibodies to Lebrikizumab | Baseline up to Week 124 (assessed at Baseline, Weeks 4, 12, 24, 36, 52, 64, 76, 92, 104, 112, and 124)
Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score | Baseline, Week 52
Minimum Serum Concentration (Cmin) of Lebrikizumab | Predose (0 hour) on Weeks 4, 12, 24, 36, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (232):
- United States (66):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Medical Research of Arizona; Allergy, Asthma & Immu, Scottsdale, Arizona
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Kern Allergy Med Clinic, Inc., Bakersfield, California
  - Allergy and Asthma Relief Experts, Granada Hills, California
  - Southern California Institute For Respiratory, Los Angeles, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Integrated Research Group Inc, Upland, California
  - Allergy & Asthma Medical Group; Clinical Research Division, Walnut Creek, California
  - Asthma & Allergy; Associates, P.C., Colorado Springs, Colorado
  - Storms Clinical Research; Institute, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Colorado Allergy & Asthma Centers, Pc, Denver, Colorado
  - Western States Clinical Research, Inc, Wheat Ridge, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Allergy Consultants PA, Boca Raton, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Georgia Pollens, Albany, Georgia
  - Brookstone Clinical Res Ctr, Columbus, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - DataQuest Medical Research, Lawrenceville, Georgia
  - Aeroallergy Research Labs, Savannah, Georgia
  - Atlanta Allergy & Asthma Clini, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Asthma & Allergy of Idaho, Twin Falls, Idaho
  - The Allergy and Asthma Center, Fort Wayne, Indiana
  - Cotton O'Neil Clinic; Stormont-Vail Hlth Care, Topeka, Kansas
  - Dr. Paul Shapero, Bangor, Maine
  - Asthma, Allergy & Sinus Center, Baltimore, Maryland
  - Chesapeake Clinical Research, Baltimore, Maryland
  - Howard County Center for Lung and Sleep, LLC, Columbia, Maryland
  - Infinity Medical Research Inc, North Dartmouth, Massachusetts
  - Clinical Research Inst, Minneapolis, Minnesota
  - Asthma and Allergy Physicians LLC, Brockton, Mississippi
  - Allergy Associates, Inc., Chesterfield, Missouri
  - Center For Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Center, L.L.C., St Louis, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - Adult Pediatric Allergy Central Jersey, Edison, New Jersey
  - Patrick V. Perin, MD, Teaneck, New Jersey
  - University of New Mexico; School of Med, Albuquerque, New Mexico
  - Winthrop Univ Hospital, Mineola, New York
  - Allergy Partners of Western NC, Asheville, North Carolina
  - Allergy & Asthma Centre of Dayton, Centerville, Ohio
  - Integrity People Services Research Company, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma Clinical Research LLC, Oklahoma City, Oklahoma
  - Vital Prospects Clin Res Pc, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Neem Research Group, Inc., Columbia, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Upstate Pharmaceutical Research; Greenville, Greenville, South Carolina
  - Future Search Clinical Trials L.P., Austin, Texas
  - Elliot J. Ginchansky, MD, PA, Dallas, Texas
  - EPIMRD, Inc. DBA Western Sky Medical Research, El Paso, Texas
  - Baylor College of Medicine; Dept of Medicine, Houston, Texas
  - Allergy & Asthma Clin Cen TX, Round Rock, Texas
  - Quality Assurance Research Ctr, San Antonio, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Allergy & Asthma Research Center, San Antonio, Texas
  - Live Oak Allergy & Asthma Clinic, San Antonio, Texas
  - Allergy Associates of Utah, Murray, Utah
  - Pulmonary Research of Albingdon, Abingdon, Virginia
  - University of Wisconsin;Allergy & Asthma Clinical Research, Madison, Wisconsin
- Argentina (5):
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - Fundacion Cidea, Buenos Aires
  - Centro Respiratorio Infantil, Rosario
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - CEMER Centro Médico de Enfermedades Respiratorias, Vicente López
- Australia (5):
  - Concord Repatriation General Hospital; Department Thoracic Medicine, Sydney, New South Wales
  - AusTrials, Brisbane, Queensland
  - Princess Alexandra Hospital, Department of Respiratory and Sleep Medicine, Brisbane, Queensland
  - Respiratory Clinical Trials Pty Ltd, Toorak Gardens, South Australia
  - The Lung Institute of Western Australia; Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (2):
  - Private Practice, Jambes
  - UZ Leuven Gasthuisberg, Leuven
- Bulgaria (10):
  - Specialized Hospital for Active Treatment for pneumo-phtysiatric diseases, Rousse
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - 5TH MHAT; Pulmonology, Sofia
  - National Multiprofile Hospital Tsar Boris III, Sofia
  - Medical Center for Specialized Outpatient Medical Care for Pulmonary Diseases, Sofia
  - SHATPD Sveta Sofia; Clin Pulmonary Diseases, Sofia
  - Alitera - Med - Medical Center EOOD, Sofia
  - Multiprofile Hospital For Active Treatment prof Kirkovich, Stara Zagora
  - Diagnostic and Consulting Centre Mladost - M OOD, Varna
  - Medical Center Tara OOD, Veliko Tarnovo
- Canada (5):
  - Cheema Research, Inc, Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Manna Research, Toronto, Ontario
  - Dr Anil Dhar Professional Medicine Corporation, Windsor, Ontario
  - Del Carpio Jaime Dr - Allergiste & Immunologue, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Thomayerova nemocnice, Praha 4 - Krc
  - Ordinace pro tuberkulozu a respiracni nemoci, Strakonice
  - KASMED, s.r.o.; Alergologie a klinicka imunologie, Tábor
- France (4):
  - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de La Croix Rousse, Lyon
  - Groupe Hospitalier Cochin St Vincent de Paul La Roche Guyon, Paris
  - Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris
- Germany (3):
  - Medaimun GmbH, Frankfurt am Main
  - Pneumologisches Forschungsinstitut, Großhansdorf
  - Praxis Dr. med. Hermann A. Trauth, Marburg
- Hungary (3):
  - Debreceni Egyetem, Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - Selye János Kórház és Rendelőintézet; Allergológiai Szakrendelés, Komárom
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center; Pulmonary Institute, Jerusalem
  - Nazareth EMMS Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
- Italy (7):
  - Azienda Ospedaliera Monaldi, Napoli, Campania
  - Azienda Ospedaliera Universitaria di Modena, Modena, Emilia-Romagna
  - Università Cattolica del Sacro Cuore UOC Allergologia- Policlinico Gemelli, Rome, Lazio
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia; S.S. Fisiopatologia Respiratoria, Pavia, Lombardy
  - P.O. Citta' Di Sesto S. Giovanni, Sesto San Giovanni, Lombardy
  - Azienda Policlinico Vittorio Emanuele; Pneumologia Riabilitativa E Allergologia, Catania, Sicily
- Japan (25):
  - Banbuntane Hotokukai Hospital, Aichi
  - Fukuoka National Hospital, Fukuoka
  - Hiroshima Allegy & Respiratory Clinic, Hiroshima
  - Ibarakihigashi National Hospital, Ibaraki
  - Uno Naikakokyukika Clinic, Isesaki-shi
  - Yokohama City University Medical Center; Neurology, Kanagawa
  - Sagamihara National Hospital, Kanagawa
  - Kumamoto Saishunso National Hospital, Koshi-shi
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Respiratory Medicine, Kyoto
  - Machida Municipal Hospital, Machida-shi
  - Hikarigaoka Spellman Hospital; Rheumatology, Miyagi
  - Nagoya Ekisaikai Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Takatsuki Red Cross Hospital; Division of Diabetes / Endocrinology / Lifestyle-Related Disease, Osaka
  - Kinki University Hospital, Osaka
  - Kishiwada City Hospital, Osaka
  - Tohoku Medical and Pharmaceutical University Wakabayashi Hospital, Sendai
  - Iwata City Hospital, Shizuoka
  - Takamatsu Municipal Hospital, Takamatsu
  - Hanzomon Hospital, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Toyama City Hospital, Toyama
- Mexico (3):
  - Centro de Investigacion Medico Biologico y Terapia Avanzada, S.C., Guadalajara
  - Unidad de Investigacion Clinica En Medicina (Udicem) S.C., Monterrey
  - Consultorio Especialidad Alergologia Pediatrica, Villahermosa
- New Zealand (4):
  - Greenlane Clinical Centre, Auckland
  - Canterbury Respiratory Research Group; Respiratory, Christchurch
  - P3 Research, Tauranga
  - Medical Research Inst. of New Zealand; Respiratory, Wellington
- Peru (9):
  - Hospital Nacional Adolfo; Guevara Velasco Essalud, Cusco
  - Hospital Nacional Luis N Saenz PNP, Lima
  - Clinica Internacional, Lima
  - ABK Reuma SRL- Medicentro BioCiencias, Lima
  - Centro de Investigación Ricardo Palma, Lima
  - Instituto Peruano de Investigacion en Ciencias Medicas, Lima
  - Clinica San Pablo, Lima
  - Clinica San Borja, Lima
  - Clinica los Andes, Miraflores
- Poland (12):
  - SP ZOZ Bienkowka- Osrodek Zdrowia w Bienkowce, Bieńnkówka
  - GRAŻYNA JASIENIAK-PINIS ATOPIA Niepubliczny Zakład Opieki Zdrowotnej Poradnie Specjalistyczne, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Specjalistyczna Poradnia Pulmonologiczna, Ostrów Wielkopolski
  - Niepubliczny Zespol Poradni Specjalistycznych PULS Poradnia Chorob Pluc i Gruzlic, Piła
  - ABC-PULMO Poradnia Chorob Pluc, Radom
  - Niepubliczny Zaklad Opieki Zdrowotnej PROFILAKTYKA Wladyslaw Pierzchala, Ruda Śląska
  - Centrum Medyczne Ogrodowa, Skierniewice
  - Alergo Medical Specjalistyczna Przychodnia Lekarska, Tarnów
  - Lexmedica, Wroclaw
  - Dobrostan Gabinety Lekarskie, Wroclaw
  - NZOZ Lekarze Specjalisci, Wroclaw
- Romania (4):
  - Spitalul Clinic de Pneumoftiziologie Leon Daniello Cluj-Napoca, Sectia Clinica Pneumologie I, Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie Palazu Mare Constanta, Palazu Mare
  - Targu Mures Clinical Emergency County Hospital, Târgu Mureş
  - Dr. Victor Babes Pneumology and Infectious Diseases Clinical Hospital, Timișoara
- Russia (13):
  - City Clinical Hospital #13, Moscow
  - I.M. Sechenov Moscow State Medical University the Ministry of Health and Social Development of RF, Moscow
  - City Clinical Hospital #2, Novosibirsk
  - Penza Regional Clinical Hospital Named After N. N. Burdenko; Therapy Department, Penza
  - Ryazan Regional Clinincal Cardiology Dispensary, Ryazan
  - Municipal Polyclinic #25, Saint Petersburg
  - St.Petersburg State Budget Healthcare Institution City Hospital of Saint Venerable Martyr Elizabeth, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - City Hospital #40 of Resort Administrative District, Saint Petersburg
  - Saratov State Medical Univ; Clinical Immun & Allerg, Saratov
  - Siberian State Medical University, Tomsk
  - Municipal Budgetery Clinical Institution of Healthcare; NA Semashko City Hospital, Yaroslavl
  - Yaroslavl State Medical Academy - Clinical Hospital #2, Yaroslavl
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Institute of Lung Diseases Vojvodina, Kamenitz
  - Clinical Hospital Centre Zemun, Zemun
- Slovakia (3):
  - Pneumo-Alergo Centrum s.r.o., Bratislava
  - ZAPA JJ Sro, Levice
  - Imunoalergologia Dzurilla s.r.o., Nitra
- South Africa (7):
  - Respiratory Research Unit, Cape Town
  - Tiervalei Trial Centre, Cape Town
  - St Augustines Hospital; Infectoilogy, Durban
  - Dr PJ Sebastian, Durban
  - Aliwal Shoal Medical Center, eMkhomazi
  - Limpopo Clinical Research Initiative; Tamboti Medical Centre, Tabazimbi
  - Clinical Projects Research, Worcester
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Seoul National University Hospital; Division of Allergy and Clinical Immunology, Seoul
  - Ewha Womans University Medical Center, Seoul
- Spain (7):
  - Complexo Hospitalario Universitario de Santiago CHUS - Hospital de Conxo, Santiago de Compostela, La Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda; Servicio de Neumología, Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Instituto de Ciencias Medicas, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala de Serveis Medics, Girona
  - Hospital Universitario la Paz; Servicio de Alergologia, Madrid
- Ukraine (13):
  - Kyiv City Tuberculosis Hospital #1; Department of Differential Diagnosis of Lung Diseases, Kyiv, Kiev Governorate
  - Municipal Institution Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - MI Dnipropetrovsk clinical association of emergency care of Dnipropetrovsk regional council, Dnipropetrovsk
  - Donetsk Municipal Treatment and Prophylactic Institution Central City Clinical Hospital #1, Donetsk
  - Municipal Institution of Health Care City Clinical Hospital #13, Kharkiv
  - SI Institute of Therapy n.a. L.T. Mala of National Academy of Medical Sciences of Ukraine, Kharkiv
  - SI National Institute of Phthisiology and Pulmonology n.a. F.G.Yanovskyi under NAMS of Ukraine, Kyiv
  - City Hospital #1, Mykolaiv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - City Clinical Hospital No.1; Therap Ukr Med Stom Acad, Poltava
  - Scientific and Research Institute of Invalid Rehabilitation of Moh of Ukraine, Vinnytsia
  - LLC Diaservis, Zaporizhzhia
  - Municipal Institution Zaporizhzhia City Multifield Clinical Hospital #9, Zaporizhzhye
- United Kingdom (4):
  - Raigmore Hospital, Inverness
  - Royal Preston Hospital, Preston
  - Royal Hallamshire Hospital; Department of Oncology, Sheffield
  - Southmead Hospital, Westbury-on-Trym, Bristol

REFERENCES:
- [Derived] Chen M, Shepard K 2nd, Yang M, Raut P, Pazwash H, Holweg CTJ, Choo E. Overlap of allergic, eosinophilic and type 2 inflammatory subtypes in moderate-to-severe asthma. Clin Exp Allergy. 2021 Apr;51(4):546-555. doi: 10.1111/cea.13790. Epub 2021 Jan 7. PMID 33217063
- [Derived] N Bauer R, Yang X, L Staton T, Olsson J, Holweg CTJ, R Arron J, Matthews JG, Choy DF. Seasonal variability of lung function and Asthma Quality of Life Questionnaire Scores in adults with uncontrolled asthma. BMJ Open Respir Res. 2019 Nov 11;6(1):e000406. doi: 10.1136/bmjresp-2019-000406. eCollection 2019. PMID 31803473
- [Derived] Hanania NA, Korenblat P, Chapman KR, Bateman ED, Kopecky P, Paggiaro P, Yokoyama A, Olsson J, Gray S, Holweg CT, Eisner M, Asare C, Fischer SK, Peng K, Putnam WS, Matthews JG. Efficacy and safety of lebrikizumab in patients with uncontrolled asthma (LAVOLTA I and LAVOLTA II): replicate, phase 3, randomised, double-blind, placebo-controlled trials. Lancet Respir Med. 2016 Oct;4(10):781-796. doi: 10.1016/S2213-2600(16)30265-X. Epub 2016 Sep 5. PMID 27616196